CLINICAL TRIAL: NCT03651219
Title: Mesylate Apatinib Combined With Irinotecan in Treatment of Recurrent Small Cell Lung Cancer: A Randomized Controlled Clinical Trial
Brief Title: Mesylate Apatinib Combined With Irinotecan in Treatment of Recurrent Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chest Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20171301
Record Dates: First submitted 2018-08-03; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Small Cell Lung Cancer
Keywords: SCLC; apatinib; Irinotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — apatinib; Irinotecan

STUDY DESIGN:
Intervention Model Description: experimental group: Irinotecan 80mg/m2 d1,d8 vi, apatinib mesylate tablets(250mg/d) po, 4-6 cycle（21d per cycle）; controlled group: Irinotecan 80mg/m2 d1,d8 vi, 4-6 cycle（21d per cycle）;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients use Apatinib Mesylate tablets combined with Irinotecan.
  Interventions: Drug: Apatinib; Drug: Irinotecan
- controlled group (Active Comparator): Patients use Irinotecan
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Apatinib — Apatinib Mmesylate tablets 250mg/d, po, there's totally 4-6 cycles(21days per cycle)
  Arms: experimental group
Drug: Irinotecan — Irinotecan 80mg/m2 d1, d8, vi, there's totally 4-6 cycles(21days per cycle)

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of apatinib mesylate tablets and chemotherapy drug Irinotecan in treatment of recurrent SCLC stage IIIB&IV patients. It is a randomized controlled clinical trial.

DETAILED DESCRIPTION:
Apatinib mesylate is a new inhibitor of VEGFR-2 tyrosine kinase targeting the intracellular ATPbinding site of the receptor.

This research needs participants satisfied following criteria:

1. Aged between 18 and 70；
2. Locally advanced/metastatic small lung cancer (IIIB/IV) confirmed by pathology with measurable lesions；
3. Patients who was treated by platinum chemotherapy drugs（including sensitive recurrency and resistant recurrency）
4. ECOG：0-2；
5. the function of primary organs is normal.
6. Patients voluntarily entered the study and signed informed consent form (ICF).

The primary goal of this research choose ORR, DCR and adverse effects as main curative effect criteria. PFS, OS and QoL as secondary curative effect criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced/metastatic small lung cancer (IIIb / IV) confirmed by pathology with measurable lesions ；
2. Patients was treated by platinum chemotherapy drugs and was diagnosed to PD；
3. ECOG：0-2；
4. Anticipated survival time more than 3 months；
5. Fertile woman must perform a pregnancy test (serum or urine) 7 days before screened, or voluntarily adopt proper methods of contraception during the observation period and 8 week after the last given apatinib. For man, surgical sterilization should be performed, or voluntarily adopt proper methods of contraception during the observation period and 8 week after the last given apatinib；
6. Patients voluntarily entered the study and signed informed consent form (ICF).
7. The function in main organs of patients is normal.

Exclusion Criteria:

1. Blend cancer type with NSCLC or else；
2. Brain MRI, CT or venography confirmed that there are brain hemorrhage symptoms;
3. MRI, CT or venography confirmed that tumor invaded big vessels;
4. Patients with uncontrollable hypertension (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg, despite optimal drug therapy).；
5. Patients with with grade Ⅱ myocardial ischemia or myocardial infarction, poor control of arrhythmias (including QTc interval male ≥ 450 ms, female ≥470 ms)；
6. Abnormal coagulation (INR>1.5 or PT>ULN+4, or APTT>1.5 ULN), bleeding tendency or receiving coagulation therapy;
7. Urine protein≥++, or urine protein in 24 hours≥1.0g;
8. Received big surgery, had bone fracture or ulcer in 4 weeks;
9. Unhealed bone fracture or wound for long time;
10. Patients with active hepatitis B virus or hepatitis C virus infection；
11. Patients who received systemic antibiotic treatment of serious infections;
12. Pregnant and lactational woman or patients do not receive contraception;
13. Patients who are prone to bleed or use anticoagulant drugs.
14. Patients who have other uncured malignant tumors.
15. Patients who experienced bleeding symptoms of clinical significance within 3 months before screening, or with confirmed bleeding tendency such as hemorrhage of digestive tract, hemorrhagic gastric ulcer, baseline occult blood in stool ++ and above, or vasculitis, etc；
16. Random 12 months before the artery/vein thrombosis events, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.；
17. Known history of hypersensitivity to apatinib or any of it components.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-09-08 (Estimated); Primary Completion 2019-08-08 (Estimated); Study Completion 2020-08-08 (Estimated)

PRIMARY OUTCOMES:
duration of treatment | two years
  time from take apatinib to withdrawal from experiment due to adverse reaction of apatinib

SECONDARY OUTCOMES:
progress free survival and overall survival | two years
  Secondary study endpoint